CLINICAL TRIAL: NCT04465669
Title: Heterogeneity of Neointimal Healing Following Biodegradable-polymer Drug-Eluting Coronary Stent Implantation
Acronym: Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Healing Stent
Record Dates: First submitted 2020-07-02; First posted 2020-07-10 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2022-10

CONDITIONS: Coronary Heart Disease; Stable Angina Pectoris; Silent Myocardial Ischemia
MeSH Terms: conditions — Coronary Disease; Angina, Stable

STUDY DESIGN:
Intervention Model Description: About 50 patients with clinical evidence of ischemic heart disease and / or a positive functional study and documented stable angina pectoris (Canadian cardiovascular society classification (CCS)1, 2, 3 or 4), or documented silent ischemia in de-novo, native, previously unstented vessel in Tyumen Cardiology Center,will be randomly assigned undergoing implantation of Orsiro stent or Resolute Integrity stent (in a 1:1 ratio).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orsiro (Active Comparator): Implantation of a Orsiro® biolimus a9 eluting coronary stent (drug-eluting stent, DES)
  Interventions: Device: Orsiro stents
- Resolute Integrity (Active Comparator): Implantation of a Resolute Integrity® zotarolimus eluting coronary stent (drug-eluting stent, DES)
  Interventions: Device: Resolute Integrity® stents

INTERVENTIONS:
Device: Orsiro stents — Percutaneous coronary intervention with implantation of either:
  a Orsiro® biolimus a9 eluting coronary stent
  Arms: Orsiro
Device: Resolute Integrity® stents — Percutaneous coronary intervention with implantation of either:
  a Resolute Integrity® zotarolimus eluting coronary stent
  Arms: Resolute Integrity

SUMMARY:
The objective of this study is a comparative evaluation of Orsiro stent and of Resolute Integrity stent in terms of the extent of neointima formation at 4 months after implantation using optical coherence tomography (OCT).

DETAILED DESCRIPTION:
About 50 patients with clinical evidence of ischemic heart disease and / or a positive functional study and documented stable angina pectoris (Canadian cardiovascular society classification (CCS)1, 2, 3 or 4), or documented silent ischemia in de-novo, native, previously unstented vessel in Tyumen Cardiology Center,will be randomly assigned undergoing implantation of Orsiro stent or Resolute Integrity stent (in a 1:1 ratio).

All of the patients will receive 12 months dual antiplatelet therapy and they will be followed (at the outpatient clinic) for up to 1 year. The follow-up visits will be conducted at 4 months (including angiographic/OCT investigation), and 1 year post percutaneous coronary intervention(PCI),in order to observe the Primary Endpoint and Secondary Endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Patients with symptoms of stable angina and/or presence of a positive functional test for ischemia;
* Patient is eligible for percutaneous coronary intervention (PCI);
* Patient has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Ethical Committee of the respective clinical site.

Exclusion Criteria:

* Target lesion involving a bifurcation with a side branch ≥2.0 mm in diameter;
* Target lesion located in the left main stem;
* Target lesion is located or supplied by an arterial or venous bypass graft;
* Lesion located very distally, difficult to be imaged by OCT;
* Co-morbidities that could interfere with completion of study procedures, or life expectancy less than 1 year;
* Participating in another investigational drug or device trial that has not completed the primary endpoint or would interfere with the endpoints of this study;
* Patient underwent target vessel revascularization with a DES;
* Patient presenting with acute myocardial infarction with ST elevation;
* Cerebrovascular accident within the past 12 months;
* Acute or chronic renal dysfunction (defined as creatinine greater than 2.0 mg/dl);
* Patient receiving oral anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Heterogeneous neointimal healing | 4 ± 1 months
  Endothelial coverage by Heterogeneous neointima of the stent struts assessed by optical coherence tomography

SECONDARY OUTCOMES:
Malapposed stent struts | 4 ± 1 months
  Percentage of malapposed stent struts by optical coherence tomography
Neointimal growth | 4 ± 1 months
  Neointimal thickness by optical coherence tomography
Angiographic reference vessel diameter | 4 ± 1 months
  Reference diameter of coronary artery by QCA
Clinical composite endpoints | 12 months
  Cardiac death/Target vessel MI/Clinically indicated TLR All death/All MI/All TVR (including TLR)
Stent Thrombosis | 12 months
  Definite stent thrombosis
Uncovered stent struts | 4 ± 1 months
  Percentage of uncovered stent struts by optical coherence tomography
Angiographic minimal lumen diameter | 4 ± 1 months
  Minimal lumen diameter of coronary artery by QCA;
Angiographic diameter stenosis | 4 ± 1 months
  Percent diameter stenosis by QCA;
Binary restenosis | 4 ± 1 months
  Binary restenosis by QCA;
Angiographic late lumen loss | 4 ± 1 months
  Late lumen loss by QCA;

CONTACTS AND LOCATIONS:
Overall Officials: Bessonov S Ivan, Principal Investigator — Tyumen Cardiology Research Center
Locations (1):
- Tyumen Cardiology Research Center, Tomsk National Research Medical Center, Russian Academy of Science, Tyumen, Russia

DOCUMENTS (1):
  • Study Protocol (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/69/NCT04465669/Prot_001.pdf